CLINICAL TRIAL: NCT00824343
Title: An Open Label, Multicenter Phase II Study to Evaluate Efficacy and Safety of P276-00 in Indian Subjects With Recurrent, Metastatic or Unresectable Locally Advanced Squamous Cell Carcinoma of Head and Neck
Brief Title: A Phase II Clinical Trial to Study the Efficacy and Safety of a New Drug P276-00 in Treatment of Recurrent and/or Locally Advanced Head and Neck Cancer
Acronym: MONARCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/21/08
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — P276-00

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single P276-00 arm (Experimental): This is a single experimental arm study
  Interventions: Drug: P276-00

INTERVENTIONS:
Drug: P276-00 — For patients to be recruited in amended protocol, P276-00 will be administered to all subjects at a dose of 144 mg/m2/day as i.v infusion in 200 ml of 5% dextrose over 30 minutes from day 1 to day 5 and from day 8 to day 12 in each 21 day cycle. Subjects will receive treatment till progression of disease or till unacceptable toxicity. All subjects will be followed up for survival status till one year of initiation of protocol treatment.

SUMMARY:
This is a single arm phase II trial to study the efficacy and safety of a Cdk inhibitor P276-00 in the treatment of squamous cell carcinoma of head and neck. Patients with recurrent or metastatic disease that is unresectable and incurable by radiation will be enrolled. Thirty eight evaluable patients need to be enrolled in the study. All patients will receive protocol treatment i.e. P276-00 as an intravenous infusion from day 1 to day 5 and from day 8 to day 12 in each 21 day cycle till progression of disease or unacceptable toxicity. Safety evaluations by means of recording vitals, physical examination and lab investigations like hematology and clinical chemistry will be undertaken at regular intervals in each cycle. Tumor measurements by spiral CT scan will be undertaken at baseline and at the end of every 2 cycles for response evaluation by RECIST criteria. All patients will be followed up for survival status till one year of cycle 1 day 1.

DETAILED DESCRIPTION:
P276-00 was administered at a dose of 185mg/m2/day from day 1 to day 5 in each 21 day cycle. The protocol was amended in July 2009. As per the amendment P276-00 will be administered at a dose of 144 mg/m2/day from day 1 to day 5 and from day 8 to day 12 in each 21 day cycle till progression of disease or unacceptable toxicity.33 patients have been recruited in version 1 protocol, 38 more evaluable patients need to be recruited in version 2 protocol. Allowing for approximately 30% drop-outs, it is estimated that, for enrolling 38 evaluable subjects in the study, approximately 54 subjects would be enrolled. As the study has already enrolled 33 subjects, the sample size for the study to accommodate for same number of subjects (38 evaluable) in the revised protocol is estimated as approximately 87 (33 + 54) subjects. Hence the total sample size (accounting for drop-outs) is 87 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than or equal to 18 years
2. Subjects with histologically or cytologically confirmed SCCHN that is recurrent and/or metastatic and judged incurable by surgery and/or radiation therapy and with zero to one line of chemotherapy for recurrent or metastatic disease at least 60 days prior to study entry.
3. Measurable disease, defined as at least one unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥10 mm by spiral computerized tomography (CT) scan or magnetic resonance imaging (MRI)
4. Tumor that is accessible to biopsy
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Life expectancy of at least three months
7. Hemoglobin ≥ 8.0 gm/dL
8. Absolute neutrophil count (ANC) ≥ 1000/mm3
9. Platelet count ≥ 50,000/mm3
10. Total bilirubin ≤1.5X institutional upper limit of normal (ULN)
11. Serum AST ≤ 3X institutional ULN
12. Serum ALT ≤ 3X institutional ULN
13. Serum creatinine ≤1.5X institutional ULN
14. Ability to understand and the willingness to sign a written informed consent document (ICD)

Exclusion Criteria:

1. Nasopharyngeal carcinoma
2. Prior treatment with P276-00 or other Cyclin dependent kinase (CDK) targeting agents
3. History of allergic reactions attributed to compounds of similar chemical composition to P276-00
4. Subjects who have received radiotherapy, chemotherapy or biologic/targeted anticancer agents within 60 days prior to Day 1 of study drug administration or have not recovered from adverse effects of any prior radiotherapy, chemotherapy or biologic/targeted agents.
5. More than one chemotherapy regimen for the recurrent or metastatic disease
6. Subjects who had received any other investigational drug within 1 month or within five half-lives of the other investigational agent, whichever is longer prior to Day 1 of study drug administration
7. Subjects with QTc > 450 msec on 12 lead standard electrocardiogram (ECG)
8. History of unstable angina or myocardial infarction or stroke within previous 6 months
9. Subjects with uncontrolled inter-current illness including, but not limited to active infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
10. Subjects known to be suffering from infection with HIV, Tuberculosis, Hepatitis C or Hepatitis B
11. Known brain metastasis
12. History of prior malignancy except for curatively treated basal cell or squamous cell carcinoma of skin, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or any other cancer for which the subject has been disease-free for at least 3 years
13. Women who are pregnant or lactating
14. Women of childbearing potential [defined as sexually mature women who have not undergone hysterectomy or who have not been naturally postmenopausal for at least 24 consecutive months (i.e. who have had menses any time in the preceding 24 consecutive months)] and men, not agreeing to use adequate contraception (e.g., hormonal or barrier method of birth control or abstinence) prior to study entry (after signing the ICD), during the period of study participation and for at least 4 weeks after withdrawal from the study, unless they are surgically sterilized
15. Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at an unacceptable risk or deems the subject not suitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Response rate | Tumor measurements to be undertaken at baseline and at the end of every 2 cycles. Response evaluation to be performed on the basis of RECIST criteria

SECONDARY OUTCOMES:
Duration of response, Progression free survival (PFS), Time to progression (TTP), PFS at one year, Overall survival (OS) at one year | Tumor measurements at the end of every 2 cycles. Follow up for survival status every 4 weeks after discontinuation of protocol treatment till one year of cycle 1 day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ajay Mehta, Principal Investigator — Director and Onco-Surgeon, Central India Cancer Research Institute, Nagpur; Dr. M S Vishveshwara, Principal Investigator — Radiation Oncologist, Bharat Hospital Institute of Oncology, Mysore; Dr. Sanjeev Misra, Principal Investigator — Oncosurgeon, Department of Surgical Oncology, CSM Medical University, Lucknow; Dr. Rejnish Kumar, Principal Investigator — Associate Professor, Regional Cancer Centre, Trivandram; Dr. Lalit Mohan Sharma, Principal Investigator — Consultant Medical Oncologist, Bhagwan Mahavir Cancer Hospital and Research Centre, Jaipur; Dr. Maheboob Basade, Principal Investigator — Medical Oncologist, Jaslok Hospital, Mumbai; Dr. Nilesh Lokeshwar, MD, DM, Principal Investigator — Medical Oncologist; Dr. Chetan Deshmukh, MD, DM, Principal Investigator — Medical Oncologist, Deenanath Mangeshkar Hospital and Research Centre, Pune, India; Dr. M Nagarajan, MD, Principal Investigator — Radiation Oncologist, V. N. Cancer Centre, GKNM Hospital, Coimbatore, India
Locations (9):
- India (9):
  - Bharath Hospital & Institute of Oncology, Mysore, Mysore, Karnataka
  - Regional Cancer Centre, Trivandrum, Kerala
  - Kashyap Nursing Home, Mumbai, Maharashtra
  - Jaslok Hospital, Mumbai, Mumbai, Maharashtra
  - Central India Cancer Research Institute,, Nagpur, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Bhagwan Mahaveer Cancer Hospital & Research Centre, Dept. Of Medical Oncology, Jaipur, Jaipur, Rajasthan
  - V. N. Cancer Centre, GKNM Hospital,, Coimbatore, Tamil Nadu
  - Dept. Of Surgical Oncology, CSM Medical University, Lucknow, Lucknow, Uttar Pradesh